CLINICAL TRIAL: NCT03539510
Title: Randomized Controlled Trial of an Interactive Website for Heart Failure Advance Care Planning
Brief Title: Effectiveness of the HF-ACP Website Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jane MacIver, Ted Rogers Nursing Professor in Cardiovascular Research, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HF-ACP website
Record Dates: First submitted 2017-07-04; First posted 2018-05-29 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure; Advance Care Planning
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: will be conducted using a single center, double-blind randomized controlled trial with 2 groups; an intervention group using the HF-ACP website and control group receiving usual care.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HF-ACP Website (Experimental): The HF-ACP website leads participants through 4 e-learning modules. Each module contains 3 core elements: (1) educational content which provides information and support to help patients complete the module (2) interactive tools for documenting their thoughts and progress and (3) motivational video clips that encourage behavior change by validating participants ambivalence, suggesting strategies to help participants complete the task and to encourage and reassure participants that they can do this.
  Interventions: Behavioral: HF-ACP Website
- Usual Care (No Intervention): The standard of care for advance care planning at our institution is the "Speak Up" booklet and the Power of Attorney workbook from the Attorney General's Office - Ontario. Patients randomized to the Control arm will be asked to register on a separate research portal where participants will have electronic access to both of the booklets and a link to the Speak Up online Interactive workbook. There is no specific information on HF or HF treatments. Participants in the control arm will be asked to complete the ACP using the interactive workbook. Participants in the control arm will not receive any additional communication from the research team about their progress.

INTERVENTIONS:
Behavioral: HF-ACP Website — Each module is broken down into weekly topics and each module takes 3-6 weeks to complete. Participants can access and review the material as often as needed as well as revisiting the information from modules they have completed.
  Arms: HF-ACP Website

SUMMARY:
This study evaluates the effectiveness of an interactive website on advance care planning for patients living with heart failure (HF-ACP website). The investigators will randomize patients to either the HF-ACP website or usual care to determine if the participants who use the HF-ACP website have higher advance care planning completion rates than participants assigned to usual care.

DETAILED DESCRIPTION:
Advance care planning is a process that supports adults at any age or stage of health to understand and share their personal values, life goals and preferences in order to prepare for future decisions regarding medical care. Public awareness campaigns to promote ACP have been taking place for about 10 years without significant improvements in ACP completion rates. Content intended for use by the general public may be too vague for those living with a chronic illness. Framing ACP within the context of a specific disease may provide the impetus for a person to engage in ACP. The investigators believe the HF-ACP website will improve patient understanding of the life-limiting nature of HF, the ACP process and the need to plan ahead to help ensure the care they receive matches their treatment preferences.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18,
* a regular patient in our clinic,
* able to read and write English,
* familiar with the use and have access to a personal computer, email and the internet.

Exclusion Criteria:

* ineligible for participation in the trial if they do not meet the inclusion criteria described above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Advance care planning completion rates | 6 months
  proportion of participants who complete the advance care planning process

SECONDARY OUTCOMES:
advance care planning knowledge | 6 months
  % improvement in knowledge of advance care planning
The 5-level European Quality of Life scale | 6 months
  The EQ-5D-5L is a generic quality of life measure that consists of a 5-item health state assessment and a visual analog scale. The dimensions represented in the 5-item assessment include: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Responses to the questions can be converted to a time tradeoff utility score from 0 (represents worst possible health) to 1.0 (represents perfect health). The visual analog scale ranges from 0-100 with higher scores representing better quality of life.
Generalized Anxiety Disorder Scale (GAD-7) | 6 months
  The GAD-7 is a 7 item self-administered screening tool for anxiety. Scores range from 0-21 with cutoffs at 5, 10, and 15 representing mild, moderate and severe anxiety, respectively.
The Readiness to Change Scale (RCS) | 6 months
  The RCS is a study-specific tool based on Prochaska's algorithm for change. It categorizes participants into one of the 5 categories of readiness. The RCS will be used to measure change for the 3 discreet behaviors: (1) identifying a SDM, (2) developing the advance care plan and (3) communicating wishes to their SDM. The RCS will be used to determine if readiness is associated with ACP completion
The Patient Health Questionnaire (PHQ-9) | 6 months
  The PHQ -9 is a 9 item self-administered scale screening tool for depression. Scores range from 0-27 with cutoffs at 5, 10, 15 and 20 representing mild, moderate, moderately severe and severe depression
The Perceived Stress Scale | 6 months
  The PSS is a 10 item self-administered scale to measure perceived stress. The scores range form 0-40 with higher scores representing greater stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Maciver, RN PhD, Principal Investigator — UHN Toronto

IPD SHARING:
Plan to Share IPD: No